CLINICAL TRIAL: NCT00209326
Title: A Randomised, Double-blind, Parallel Group, Dose-ranging, Placebo-controlled, Multi-centre, Proof of Concept Study Assessing the Effect of Four Different Single Bolus Intravenous Doses of FE200440 (0.3, 1, 3, 10 mg) and Placebo on Stopping Preterm Labour and Uterine Contractions in Pregnant Women With Advanced Gestational Age
Brief Title: A Proof of Concept Study Assessing the Effect of Four Different Single Bolus Intravenous Doses of FE200440 and Placebo on Stopping Preterm Labor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE200440 CS004
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Labor, Premature; Premature Birth
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

INTERVENTIONS:
Drug: FE200440

SUMMARY:
• To determine the effects of four different single bolus doses of FE200440 administered intravenously on stopping preterm labour compared to placebo in pregnant women with advanced gestational age

DETAILED DESCRIPTION:
* To determine the effects of four different single bolus doses of FE200440 administered intravenously on stopping preterm labour compared to placebo in pregnant women with advanced gestational age
* To establish the effects of four different single bolus doses of FE200440 administered intravenously on uterine contractions compared to placebo
* To evaluate the effects of four different single bolus doses of FE200440 administered intravenously on labour progression compared to placebo
* To establish the dose-response curve of single bolus doses of FE200440 administered intravenously in terms of time to delivery, uterine contractions and labour progression
* To determine the duration of action of four different single bolus doses of FE200440 administered intravenously in terms of time to delivery, uterine contractions and labour progression
* To establish the pharmacokinetic parameters of FE200440 after single bolus intravenous administration
* To determine the relation between plasma concentrations of FE200440 and uterine contractions and labour progression
* To compare the maternal, fetal and infant safety profile after intravenous administration of four different single bolus doses of FE200440 and placebo
* To evaluate the impact of four different single bolus doses of FE200440 administered intravenously on delivery outcome, postpartum events and lactation

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form, prior to screening evaluations
2. Mother and fetus in good general health
3. Pregnant women age ≥ 18 years
4. Gestational age (verified by early ultrasound or if an ultrasound is not available by Last Menstrual Period) between 34 weeks + 0 days and 35 weeks + 6 days (both days inclusive)
5. At randomisation, there must be 6 or more uterine contractions of at least 30 seconds duration during a 30 minutes interval
6. At randomisation, the cervical length must be ≤ 15 mm (by transvaginal ultrasound)
7. At randomisation, the cervical dilatation must be >1 cm and <4 cm (by vaginal examination

Exclusion Criteria:

1. Contraindications for the mother or the fetus to stop labour, including

   * clinical suspicion of abruptio placenta
   * known or suspected infection (e.g. urinary tract infection, chorioamnionitis)
2. Controlled or uncontrolled diabetes mellitus (pre-gestational or gestational)
3. Eclampsia or severe preeclampsia in the current pregnancy
4. Previous major uterine surgery (e.g. myomectomy for leiomyomas), congenital uterine abnormalities, large leiomyomas, or retained intrauterine device
5. Rupture of membrane in the current pregnancy
6. Placenta praevia in the current pregnancy
7. a)
8. Oligohydramnios or polyhydramnios in the current pregnancy defined as amniotic fluid index (AFI) below 7.2 cm or above 27.8 cm
9. Fetal weight (based on ultrasound) outside the ± 2SD limits provided in Appendix B
10. Use of cervical cerclage in the current pregnancy
11. Current multiple pregnancy
12. Fetal death in utero in previous or current pregnancy
13. Fetus with known or suspected abnormal karyotype or major malformations in the current pregnancy
14. Abnormal fetal heart rate which the Investigator judges to reflect fetal distress
15. Treatment with nifedipine, non-steroidal anti-inflammatory agents (NSAIDs) or intravenously administered magnesium sulphate for contractions during the current pregnancy or treatment with beta-mimetics, atosiban or progesterone within the last 7 days prior to randomisation
16. Treatment with anticoagulation or fibrinolytic therapies prior to screening, or known or suspected or past history of thromboembolic disorders
17. Known, suspected or past history of hypocoagulability or coagulation deficiency conditions
18. Known or suspected hemoglobinopathies
19. Use of any investigational drug during the current pregnancy
20. Known, suspected or past history (last 12 months) of alcohol or drug abuse
21. Known hypersensitivity to the active ingredient or to any of its excipients

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2003-11; Primary Completion 2006-07 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (17):
- Belgium (3):
  - ULB Erasme Hospital Gynecology, Route de Lennik 808, Brussels
  - CHR Citadelle, Boulevard du 12iede Ligne 1, Liège
  - AZ Heilig Hart Gynecology, Kliniekstraat 44, Tienen
- Czechia (6):
  - Gynekologicko-porodnicka klinika Fakultni nemocnice Brno, Obilni trh 11, Brno
  - Gynekologicko-porodnicke oddeleni nemocnice Jihlava, Vrchlickeho 59, Jihlava
  - Gynekologicka-porodnicka klinika Fakultni nemocnice, Capkovo namesti 1, Pilsen
  - Gynekologicko-porodnicka klinika 1. LF UK a VFN v Praze, Apolinarska 18, Prague
  - Gynekologicko-porodnicka klinika Fakultni nemocnice Motol, V uvalu 84, Prague
  - Gynekologicko.porodnicke oddeleni, Socialni pece 12A, Ústí nad Labem
- Finland (3):
  - Kuopio University Hopital, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Kiinamyllynkatu 4-6, Turku
- Lithuania (2):
  - Kaunas Medical University Clinics, Eiveniu 2, Kaunas
  - Vilnius University, Antakalnio 57, Vilnius
- Zaklad Patofizjologii Ciazy AM w Bialymstoku, M.C. Sklodowskiej 24a, Bialystok, Poland
- Romania (2):
  - Spitalul Clinic de Urgenta "Elias", Nr. 17, Str. Marasti, sector 1, Bucharest
  - Spitalul Clinic Judetean Cluj-Napoca Ginecologie No. 1, Clinica Nr. 1 Ginecologie Nr. 3-5, Str. Clinicilor, Cluj-Napoca